CLINICAL TRIAL: NCT00183287
Title: Clinical, Virologic, and Immunologic Evaluation and Monitoring of Patients With Known or Suspected HIV Infection
Brief Title: Long Term Follow-Up of HIV Infected Patients Who Have Previously Participated in HIV Clinical Trials
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRP 020; 11754 (Registry Identifier: DAIDS ES Registry ID)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection

SUMMARY:
The purpose of this study is to monitor the progression of HIV infection and HIV-related disease processes in patients who have previously participated in HIV clinical trials.

DETAILED DESCRIPTION:
Since 1982, the National Institute of Allergy and Infectious Diseases (NIAID) has been conducting numerous clinical trials on patients infected with HIV-1. Unfortunately, once clinical studies have closed or participants have reached a study endpoint, no additional follow-up data are collected regarding progression of HIV infection and development of HIV-related complications in these study participants. This study will collect long-term data for participants of previous NIAID-sponsored clinical trials to study HIV-related disease processes and complications, benefits and toxicities of investigational medications and vaccines, and medical management of participants with known or suspected HIV infection.

Study visits will occur every 6 months. A physical exam, blood collection, and medical history will occur at all visits. Depending on the need of participants, additional laboratory and diagnostic tests will be performed, and standard medical care will be provided.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Previously participated in a NIAID-funded clinical trial studying HIV disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected individuals who have previously participated in NIAID-funded HIV clinical trials
Sampling Method: Non-Probability Sample
Enrollment: 150
Dates: Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn M. Mican, MD, Principal Investigator — Laboratory of Immunoregulation (LIR), NIAID